

School of Psychological Sciences 1400 East Hanna Avenue Indianapolis, Indiana 46227

(317) 788-3353 Fax: (317) 788-2120 http://psych.uindy.edu

Study Title: Client-directed cognitive processing therapy

Document Date: 3/23/2018

NCT02684994



School of Psychological Sciences 1400 East Hanna Avenue Indianapolis, Indiana 46227 (317) 788-3353 Fax: (317) 788-2120 http://psych.uindy.edu

Potential participants will contact the research team in response to recruitment materials and will leave a message expressing interest in the study. A research team member will return the call and conduct an initial phone screen to assess initial eligibility. If the potential participant meets initial criteria, their contact information will be passed along to a research team member to call and schedule the pretreatment assessment appointment. If the potential participant does not meet criteria, they will not proceed with the study. A list of local referrals will be mailed.

The pre-treatment assessment appointment will begin with obtaining informed consent. Next, the assessment will include 4-5 semi-structured clinical interviews. The first interview assesses posttraumatic stress disorder symptoms. The second assesses other psychological disorders. The third obtains more information about the participant's trauma history. The fourth assesses sex trafficking experiences. The optional fifth interview will only be given to people who report sex trafficking experiences. Following completion of the clinical interviews, the participant will complete self-report questionnaires assessing additional psychological symptoms, potential vulnerability factors for PTSD, and measures of functioning. If the participant is eligible for participation in the study, the participant will then be assigned to a clinician. If the participant is not eligible, then they will be provided with a list of local resources. Participants will receive a \$25 gift card for participating in the in-person assessment.

Once assigned to a clinician, the clinician will schedule the first treatment session. Treatment will primarily follow the protocol for the manualized treatment cognitive processing therapy. Treatment will include twelve 50 minute sessions which can be attended once or twice a week. The treatment protocol will be split into 4 sections [1) traditional session 1-3, 2) traditional sessions 4 & 5, 3) traditional sessions 6 & 7, and 4) traditional sessions 8 - 12]. All clients will complete the standard introduction portion (traditional sessions 1-3). At the end of session 3, clients will choose to either continue in the standard protocol manner (and complete traditional sessions 4 and 5) or begin the cognitive restructuring portion (traditional sessions 6 & 7). If the client chose to do 4 and 5 first, then the participant will complete 6 & 7 and then the topic module sessions. If the participant chose to complete 6 & 7 first, then they will be given the choice to complete the modules (traditional sessions 8 - 12) or to complete the narrative (traditional 4 & 5). Finally, the participant will complete the remaining section. Since the cognitive only version of CPT has been demonstrated to be as effective as the full CPT protocol, participants will not be required to complete the narrative (traditional sessions 4 & 5).

Approximately 2 weeks following treatment completion, or around the time treatment completion would be anticipated if the participant drops out of treatment, the participant will complete an in person post-treatment assessment. The post-treatment assessment will include many, but not all, of the same measures as the pre-treatment. The post-treatment assessment will include two semistructured interviews along with self-report measures. The participant will be given a \$25 gift card for completion of the in-person post-treatment assessment.

Finally, three months following the post-treatment assessment, a follow-up phone assessment will be scheduled. This assessment will only include two semi-structured interviews and will be conducted over the phone. The treatment team will attempt to get assessment data for treatment drop-outs as well as completers.

All protocol interactions with participants will be conducted by either a co-investigator or the PI. All data in the current study will be written onto measures either by the research team or the participant. Data will be entered into SPSS dataset(s). However, no identifiable information will be included in the dataset.



School of Psychological Sciences 1400 East Hanna Avenue Indianapolis, Indiana 46227

(317) 788-3353 Fax: (317) 788-2120 http://psych.uindy.edu

Statistical Analysis Plan

Analyses will be examined using repeated measures ANOVAs with CAPS scores as the within subjects variable. Analyses will be examined for both treatment completers and intent to treat sample. Last observation carried forward procedures will be used for the intent to treat sample. Potential covariates, including demographics and trauma type will be examined and included if relevant.